CLINICAL TRIAL: NCT04074005
Title: Incidence and Factors Involving Cesarean Delivery After Epidural Analgesia for Labor
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 020/2562 (EC4)
Record Dates: First submitted 2019-05-04; First posted 2019-08-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section; Epidural; Anesthesia
Keywords: Epidural analgesia; Labor pain; Cesarean section rate
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rate of cesarean delivery after epidural analgesia for labor has not been reported in our institute. The aim of this study is to elucidate incidence of cesarean delivery in parturient whom received epidural analgesia. Besides, factors associated with the rate of cesarean delivery were studied.

DETAILED DESCRIPTION:
Epidural analgesia with local anesthetic and opioid is the efficiently good method to relieve labor pain comparing with intravenous opioid analgesic. Many literatures reported effects epidural analgesia for labor eg. prolonging the duration of second stage of labor, increasing the rate of instrumental delivery: vacuum extraction and forceps assisting labor. Some papers revealed the increasing in the rate of cesarean delivery. The main reason is assume to be a failure to progress labor after epidural analgesia. However, the recent report from Cochrane database systematic review showed no relation of epidural analgesia for labor and the increasing in the rate of cesarean delivery. Various factors that may involve in the increasing in the rate of cesarean delivery including the dilatation of cervix at the time of insertion of epidural catheter, nulliparous, size of the fetus or motor weakness after receiving epidural medication.

The rate of cesarean delivery after epidural analgesia for labor has not been reported in our institute. The aim of this study is to elucidate incidence of cesarean delivery in parturient whom received epidural analgesia. Besides, factors associated with the rate of cesarean delivery were studied.

ELIGIBILITY:
Inclusion Criteria:

* Age>,= 18 years
* Accept epidural analgesia for labor
* ASA classification I-II

Exclusion Criteria:

* Unable to communicate Thai

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women whom admitted in labor ward for delivering baby as well as accept to receive epidural analgesia for labor
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of cesarean delivery after epidural analgesia for labor | From epidural catheter insertion to delivery
  Rate of cesarean delivery after patients receive epidural analgesia for relieve labor pain

SECONDARY OUTCOMES:
Factors affecting rate of cesarean delivery after epidural analgesia for labor | at the time epidural catheter insertion
  cervical dilatation before insertion epidural catheter (cm.)
Efficacy of epidural analgesia for labor | before and after epidural catheter insertion
  pain score (verbal rating scale pain score)
Side effects of epidural analgesia for labor: nausea and vomiting | From epidural catheter insertion to delivery
  nausea and vomiting (rating by patients: 0= no symptom, 1= nausea 2= vomiting)
Side effects of epidural analgesia for labor: pruritus | From epidural catheter insertion to delivery
  pruritus (0=no, 1=yes)
Side effects of epidural analgesia for labor: numbness of legs | From epidural catheter insertion to delivery
  numbness of legs (0=no, 1=yes)
Side effects of epidural analgesia for labor: motor weakness | From epidural catheter insertion to delivery
  Rate motor weakness by Bromage score

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nivatpumin P, Triyasunant N, Visalyaputra S, Lertbunnaphong T, Saenyasiri N. Incidence and associated factors of cesarean delivery following epidural analgesia for labor: A prospective cohort study at a Thai university hospital. Midwifery. 2025 Sep;148:104501. doi: 10.1016/j.midw.2025.104501. Epub 2025 Jun 24. PMID 40609139